CLINICAL TRIAL: NCT04311697
Title: ZYESAMI (Aviptadil) for the Treatment of Critical COVID-19 With Respiratory Failure
Brief Title: Intravenous Aviptadil for Critical COVID-19 With Respiratory Failure
Acronym: COVID-AIV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID-AIV
Expanded Access: NCT04453839 (No longer available)
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2021-09

CONDITIONS: Critical COVID-19 With Respiratory Failure; Acute Respiratory Distress Syndrome (ARDS); Corona Virus Infection; Acute Lung Injury
Keywords: COVID-19; ARDS; Aviptadil; Acute Respiratory Distress Syndrome; Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections; Acute Lung Injury; COVID-19; Respiratory Insufficiency | interventions — Standard of Care; aviptadil

STUDY DESIGN:
Intervention Model Description: Multicenter trial, initially conducted at a single center with a safety/futility assessment following enrollment of 30 patients, expanded to 196 total patients at 12 study sites
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, placebo-controlled trial with identical drug and placebo infusion bags
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aviptadil IV in escalating doses + standard of care (Experimental): Patients will be administered Aviptadil IV in escalating doses of 50 pmol, 100 pmol, 150 pmol/kg/hr
  Interventions: Drug: Aviptadil by intravenous infusion + standard of care
- Placebo + standard of care (Experimental): Patients will first be treated with placebo infusion + maximal intensive care
  Interventions: Drug: Normal Saline Infusion + standard of care

INTERVENTIONS:
Drug: Aviptadil by intravenous infusion + standard of care — Aviptadil by intravenous infusion + standard of care (SOC). SOC is defined not to include extracorporeal mechanical oxygenation. Those requiring ECMO will be withdrawn from the study as treatment failures.
  Other Names: ZYESAMI (aviptadil) +SOC
  Arms: Aviptadil IV in escalating doses + standard of care
Drug: Normal Saline Infusion + standard of care — Saline by intravenous infusion + standard of care (SOC). SOC is defined not to include extracorporeal mechanical oxygenation. Those requiring ECMO will be withdrawn from the study as treatment failures.
  Other Names: Placebo+SOC
  Arms: Placebo + standard of care

SUMMARY:
Novel Corona Virus (SARS-CoV-2) is known to cause Respiratory Failure, which is the hallmark of Acute COVID-19, as defined by the new NIH/FDA classification. Approximately 50% of those who develop Critical COVID-19 die, despite intensive care and mechanical ventilation. Patients with Critical COVID-19 and respiratory failure, currently treated with high flow nasal oxygen, non-invasive ventilation or mechanical ventilation will be treated with ZYESAMI (aviptadil), a synthetic form of Human Vasoactive Intestinal Polypeptide (VIP) plus maximal intensive care vs. placebo + maximal intensive care. Patients will be randomized to intravenous Aviptadil will receive escalating doses from 50 -150 pmol/kg/hr over 12 hours.

DETAILED DESCRIPTION:
Acute Lung Injury, which triggers Critical COVID-19 is a known lethal complication of Corona Virus (SARS-CoV-2) infection. Conventional medical therapy, including intensive care and respiratory support is associated with an 80% mortality. Aviptadil, a synthetic form of Human Vasoactive Intestinal Polypeptide (VIP) has been awarded FDA Orphan Drug Designation for the treatment of ARDS and admitted to the FDA CoronaVirus Technology Accelerator Program.

VIP binds to VPAC1 receptors on the pulmonary Alveolar Type II (ATII) cell. ATII cells comprise only 5% of lung epithelial cells but are critical for oxygen transfer, surfactant production, and maintenance of Alveolar Type 1 cells. 70% of VIP binds to this receptor. The Type II cell is also the cell selectively attacked by the SARS-CoV-2 virus via the ACE2 surface receptor.

Nonclinical studies demonstrate that VIP is highly concentrated in the lung and specifically bound to the ATII cell, where it prevents NMDA-induced caspase-3 activation in the lung, inhibits IL6 and TNFa production, protects against HCl-induced pulmonary edema, and upregulates surfactant production, These and other effects have been observed in numerous animal model systems of lung injury in mice, rats, guinea pigs, sheep, swine, and dogs. In these models, Aviptadil restores barrier function at the endothelial/alveolar interface and thereby protects the lung and other organs from failure.

Aviptadil ihas a demonstrated 20 year history of safety in phase 2 trials for Sarcoid, Pulmonary Fibrosis, Bronchospasm, and a phase I trial in ARDS. In that phase I trial, 8 patients with severe ARDS on mechanical ventilation were treated with ascending doses of VIP. Seven of the 8 patients were successfully extubated and were alive at the five day timepoint. Six left the hospital and one died of an unrelated cardiac event.

Five phase 2 trials of aviptadil have been conducted under European regulatory authority. Numerous healthy volunteer studies have shown that i.v. infusion of Aviptadil is well tolerated with few adverse effects including alterations in blood pressure, heart rate, or ECG. In addition to published studies of human use, Aviptadil has been used on a compounded basis in certain ICUs for many years in the belief that it preserves life and restores function in pulmonary hypertension, ARDS, and Acute Lung Injury (ALI).

In this study, patients who are hospitalized for Critical COVID-19 infection with respiratory failure will be randomly allocated to Aviptadil administered by intravenous infusion in addition to maximal intensive care vs. maximal intensive care alone. Primary endpoints will be improvement in blood oxygenation and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Critical COVID-19 with respiratory failure
* Physician determination that patient is on maximal conventional medical therapy

Exclusion Criteria:

1. Pregnancy (pregnant women may apply for open label treatment under compassionate care IND
2. Age <18 years
3. Mechanical ventilation for more than 7 days in primary cohort. Mechanical ventilation>21 days in the exploratory cohort
4. Mean Arterial Pressure < 65 mm Hg with use of pressor per ICU protocol
5. Irreversible condition (other than COVID-19) with projected fatal course
6. ECMO
7. Current or recent (within 30 d) enrollment in another investigational trial of anti-IL6 drug;
8. Active diagnosis of Acquired immune deficiency syndrome;
9. Transplant patients currently immunosuppressed;
10. Chemotherapy-induced neutropenia (granulocyte count <1000/mm3);
11. Cardiogenic shock; congestive heart failure - NYHA Class 3 or 4;
12. Recent myocardial infarction - within last 6 months and troponin > 0.5
13. Anuria (urine output < 50 ml/d) or other signs of multi-organ failure
14. Severe liver disease with portal hypertension;
15. Recent stroke or head trauma within last 12 months
16. Increased intracranial pressure, or other serious neurologic disorder;
17. Liquid Diarrhea more than 3x/day; defined as more than 3 non-bloody watery stools within a 24-hour period, requiring additional fluid and electrolyte supplementation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Javitt, MD, MPH, Study Chair — NeuroRx, Inc.
Locations (10):
- United States (10):
  - St. Jude Medical Center, Fullerton, California
  - University of California - Irvine, Irvine, California
  - Miller School of Medicine / University of Miami Medical Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - University of Louisville Hospital, Louisville, Kentucky
  - Heartland/Mosaic Health, Saint Joseph, Missouri
  - Hendrick Health, Abilene, Texas
  - Texas Health Harris Methodist Hospital, Fort Worth, Texas
  - Texas Health Hospital Frisco, Frisco, Texas
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NeuroRx will share study protocol and statistical analysis plan upon request by qualified researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Currently available
Access Criteria: Public access

REFERENCES:
- [Derived] Youssef JG, Lavin P, Schoenfeld DA, Lee RA, Lenhardt R, Park DJ, Fernandez JP, Morganroth ML, Javitt JC, Jayaweera D. The Use of IV Vasoactive Intestinal Peptide (Aviptadil) in Patients With Critical COVID-19 Respiratory Failure: Results of a 60-Day Randomized Controlled Trial. Crit Care Med. 2022 Nov 1;50(11):1545-1554. doi: 10.1097/CCM.0000000000005660. Epub 2022 Aug 29. PMID 36044317

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care
Started | 136 | 67
Completed | 85 | 35
Not Completed | 51 | 32

BASELINE CHARACTERISTICS:
Population: Please note that 5 patients in Aviptadil group were randomized but did not receive Investigational Product. and 2 patients in placebo group were randomized but did not receive treatment - numbers reflect those receiving investigational product
Groups:
- Total: Total of all reporting groups
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care | Total
Number analyzed (Participants) | 131 | 65 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 5 patients in aviptadil group and 2 patients in placebo group were randomized but not treated.
  years | 60.1 (12.61) | 62.7 (12.11) | 61.0 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 patients in aviptadil group and 2 patients in placebo group were randomized but not treated.
  Participants
    Female | 46 | 15 | 61
    Male | 85 | 50 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 5 patients in aviptadil group and 2 patients in placebo group were randomized but not treated.
  Participants
    Hispanic or Latino | 66 | 39 | 105
    Not Hispanic or Latino | 65 | 26 | 91
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 5 patients in aviptadil group and 2 patients in placebo group were randomized but not treated.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 7 | 1 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 10 | 5 | 15
    White | 110 | 57 | 167
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 131 | 65 | 196

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Respiratory Failure (Alive and Free of Respiratory Failure)
Description: Participant is Alive and Free of Respiratory Failure (without subsequent relapse over 7 days) determined as no longer requiring acute care or more than low flow oxygen
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 131 | 65
Participants | 72 | 33

2. Secondary Outcome: Number of Participants Alive at Day 60
Description: Survival probability on logistic regression through day 60
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 131 | 65
Participants | 85 | 35

3. Secondary Outcome: Number of Participants Achieving a Score of 6-8 on NIAID Ordinal Score Through Day 60
Description: Achievement of score 6-8 on NIAID Ordinal Scale through day 60 The NIAID score is the patient's status on the following 8-point scale:1)Death2)Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO),3)Hospitalized, on non-invasive ventilation or high flow oxygen devices4)Hospitalized, requiring supplemental oxygen5)Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)6)Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care7)Not hospitalized, limitation on activities and/or requiring home oxygen8)Not hospitalized, no limitations on activities-- a lower NIAID score is a worse outcome.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 131 | 65
Participants | 76 | 35

4. Secondary Outcome: Oxygenation Index as Measured by PaO2:FiO2 Ratio
Description: oxygenation index (also known as Respiratory Distress Ratio) as measured by PaO2:FiO2 ratio (Respiratory Distress while on mechanical ventilation). RDR: PaO2:FiO2 represents an intermediate clinical endpoint that is known to be predictive of survival. RDR can only be measured in patients on mechanical ventilation because of its reliance on arterial blood gas measurements that are not routinely collected in non-intubated patients. A higher score indicates a better clinical outcome.
Time Frame: Day 7
Population: only patients with observations were analyzed
Measure: Mean (Standard Deviation); unit: PaO2:FiO2 ratio
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 65 | 33
PaO2:FiO2 ratio | 139.2 (77.0) | 116.2 (41.77)

5. Other Pre Specified Outcome: Change in IL-6
Description: Change in IL-6, an inflammatory marker
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: IL-6 picogram/mL
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 38 | 18
IL-6 picogram/mL | 19.8 (39.9) | 23.5 (39.7)

ADVERSE EVENTS:
Time Frame: AEs were collected from administration of informed consent through the subject's hospital discharge. Any ongoing AE was followed through 60 days.
Description: Note: The numbers of patients for the PTs in a SOC may not add up to the number of patients for the SOC because patients with multiple PTs in the same SOC were counted only once. For similar reasons, the sum of the numbers of patients for the SOCs may not be the same as the number of patients with any SAE.
Arm/Group | Aviptadil IV in Escalating Doses + Standard of Care | Placebo + Standard of Care
All-Cause Mortality (participants affected / at risk) | 46/131 | 30/65
Serious Adverse Events (participants affected / at risk) | 58/131 | 32/65
Other Adverse Events (participants affected / at risk) | 102/131 | 49/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aviptadil IV in Escalating Doses + Standard of Care (N=131) | Placebo + Standard of Care (N=65)
blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
cardiac arrest (Cardiac disorders) | 5 (5) | 2 (2)
cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
pulseless electrical activity (Cardiac disorders) | 5 (5) | 2 (2)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
multiple organ dysfunction syndrome (General disorders) | 8 (8) | 9 (9)
hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 22 (22) | 10 (10)
diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
klebsiella infection (Infections and infestations) | 2 (2) | 0 (0)
pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
pneumonia infection (Infections and infestations) | 2 (2) | 0 (0)
sepsis (Infections and infestations) | 3 (3) | 1 (1)
septic shock (Infections and infestations) | 5 (5) | 3 (3)
oxygen consumption increased (Investigations) | 2 (2) | 0 (0)
oxygen saturation decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
pulse absent (Investigations) | 1 (1) | 0 (0)
hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
brain oedema (Nervous system disorders) | 0 (0) | 2 (3)
cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
superior sagittal sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 7 (7) | 5 (6)
renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 8 (8)
respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 3 (3) | 2 (2)
hypotensive crisis (Vascular disorders) | 0 (0) | 1 (1)
shock (Vascular disorders) | 1 (1) | 0 (0)
shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aviptadil IV in Escalating Doses + Standard of Care (N=131) | Placebo + Standard of Care (N=65)
anaemia (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
leukocytosis (Blood and lymphatic system disorders) | 8 (8) | 5 (5)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
atrial fibrillation (Cardiac disorders) | 15 (18) | 3 (3)
bradycardia (Cardiac disorders) | 9 (9) | 3 (4)
cardiac arrest (Cardiac disorders) | 5 (5) | 3 (3)
pulseless electrical activity (Cardiac disorders) | 5 (5) | 2 (2)
sinus arrest (Cardiac disorders) | 0 (0) | 2 (2)
sinus bradycardia (Cardiac disorders) | 3 (3) | 2 (2)
sinus tachycardia (Cardiac disorders) | 4 (5) | 0 (0)
tachycardia (Cardiac disorders) | 5 (7) | 1 (1)
ventricular tachycardia (Cardiac disorders) | 4 (6) | 5 (5)
constipation (Gastrointestinal disorders) | 9 (9) | 7 (7)
diarrhoea (Gastrointestinal disorders) | 43 (48) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
multiple organ dysfunction syndrome (General disorders) | 9 (9) | 9 (9)
oedema peripheral (General disorders) | 3 (3) | 1 (1)
pyrexia (General disorders) | 5 (5) | 1 (1)
aspergillus infection (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 22 (22) | 10 (10)
cytomegalovirus infection (Infections and infestations) | 0 (0) | 2 (2)
herpes simplex (Infections and infestations) | 1 (1) | 2 (2)
sepsis (Infections and infestations) | 4 (4) | 1 (1)
septic shock (Infections and infestations) | 6 (6) | 4 (4)
infusion related reaction (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
mechanical ventilation complication (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
alanine aminotransferase increased (Investigations) | 4 (4) | 4 (4)
aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1)
base excess increased (Investigations) | 1 (1) | 3 (3)
blood bicarbonate increased (Investigations) | 1 (1) | 3 (3)
blood creatinine increased (Investigations) | 3 (3) | 1 (1)
blood lactic acid increased (Investigations) | 3 (3) | 2 (2)
blood pH increased (Investigations) | 2 (2) | 2 (2)
haematocrit decreased (Investigations) | 1 (1) | 2 (2)
mean cell haemoglobin increased (Investigations) | 3 (3) | 0 (0)
metamyelocyte count increased (Investigations) | 1 (1) | 2 (2)
monocyte count increased (Investigations) | 2 (2) | 3 (3)
myelocyte count increased (Investigations) | 2 (2) | 2 (2)
neutrophil count increased (Investigations) | 3 (3) | 0 (0)
oxygen saturation decreased (Investigations) | 4 (6) | 3 (4)
PCO2 decreased (Investigations) | 2 (2) | 2 (2)
PO2 decreased (Investigations) | 0 (0) | 2 (2)
protein total decreased (Investigations) | 4 (4) | 2 (2)
urine output decreased (Investigations) | 4 (4) | 1 (1)
white blood cell count increased (Investigations) | 3 (3) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
fluid overload (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
hyperkalaemia (Metabolism and nutrition disorders) | 16 (16) | 4 (4)
hypernatraemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
metabolic acidosis (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
dizziness (Nervous system disorders) | 3 (3) | 0 (0)
encephalopathy (Nervous system disorders) | 4 (4) | 2 (2)
headache (Nervous system disorders) | 0 (0) | 2 (2)
toxic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
agitation (Psychiatric disorders) | 3 (3) | 2 (2)
anxiety (Psychiatric disorders) | 6 (6) | 3 (3)
confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
depression (Psychiatric disorders) | 0 (0) | 2 (2)
insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
restlessness (Psychiatric disorders) | 6 (6) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 31 (32) | 13 (14)
anuria (Renal and urinary disorders) | 3 (3) | 1 (1)
azotaemia (Renal and urinary disorders) | 4 (4) | 1 (1)
renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3)
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (8)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 9 (9)
tachypnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (6)
deep vein thrombosis (Vascular disorders) | 17 (19) | 9 (10)
flushing (Vascular disorders) | 13 (19) | 2 (2)
hypertension (Vascular disorders) | 3 (3) | 1 (1)
hypotension (Vascular disorders) | 34 (45) | 14 (19)
hypotensive crisis (Vascular disorders) | 0 (0) | 2 (2)
shock (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT04311697/Prot_SAP_000.pdf